CLINICAL TRIAL: NCT03910218
Title: Come As You Are - Assessing the Efficacy of a Nurse Case Management HIV Prevention and Care Intervention Among Homeless Youth
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Collaborators: National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Principal Investigator, Diane Santa Maria, Associate Professor, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: HSC-SN-18-0993
Record Dates: First submitted 2019-04-08; First posted 2019-04-10 (Actual); Results first posted 2025-06-26 (Actual); Last update posted 2025-06-26 (Actual); Status verified 2025-06

CONDITIONS: Behavior, Risk
Keywords: HIV prevention; homeless
MeSH Terms: conditions — Risk-Taking

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- NCM4HIV (Experimental): Participant will receive NCM4HIV intervention which includes Personalized HIV prevention education, behavior goal-setting,behavioral self-monitoring,Pre exposure prophylaxis (PrEP) eligibility screening,PrEP/non occupational post exposure prophylaxis(nPEP)services (labs, medication), healthcare planning/coordination, Motivational Interviewing (MI) counseling approach, assisting with cognitive appraisals (clarifying misconceptions),promoting health seeking and coping behaviors that incorporate the situational, personal, social, and resource needs affecting health
  Interventions: Behavioral: NCM4HIV
- Usual care (Placebo Comparator): Participants will receive the usual care which includes Housing, food, and clothing needs,health assessment, basic healthcare, limited anticipatory guidance, mental health counseling,substance use treatment referrals,PrEP/nPEP referrals
  Interventions: Behavioral: Usual Care

INTERVENTIONS:
Behavioral: NCM4HIV — Participant will receive NCM4HIV intervention which includes Personalized HIV prevention education, behavior goal-setting,behavioral self-monitoring, PrEP eligibility screening,PrEP/nPEP services (labs, medication), healthcare planning/coordination, MI counseling approach, assisting with cognitive appraisals (clarifying misconceptions),promoting health seeking and coping behaviors that incorporate the situational, personal, social, and resource needs affecting health
  Arms: NCM4HIV
Behavioral: Usual Care — Participant will receive usual care which includes Housing, food, and clothing needs,health assessment, basic healthcare, limited anticipatory guidance, mental health counseling, substance use treatment referrals, PrEP/nPEP referrals
  Arms: Usual care

SUMMARY:
The purpose of this study is to to determine the efficacy of the Nurse Case Management HIV (NCM4HIV) intervention on HIV prevention compared to usual care among Youth Experiencing Homelessness (YEH).

ELIGIBILITY:
Inclusion Criteria

* youth engaged in high-risk sexual activity or intravenous drug use
* speak English
* homeless
* not planning to move out of the metro area during the study

Exclusion Criteria:

* youth with very low literacy
* severe acute mental symptoms

Ages: 16 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 474 (Actual)
Dates: Start 2019-11-11 (Actual); Primary Completion 2024-04-03 (Actual); Study Completion 2024-04-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Diane Santa Maria, DrPH, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- The University of Texas Health Science Center at Houston, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Maria DS, Nyamathi A, Lightfoot M, Paul M, Quadri Y, Padhye N, Businelle M, Fernandez-Sanchez H, Jones JT. Results of a Randomized Wait-List Controlled Trial of CAYA: A Nurse Case Management HIV Prevention Intervention for Youth Experiencing Homelessness. AIDS Behav. 2025 Feb;29(2):613-625. doi: 10.1007/s10461-024-04544-3. Epub 2024 Nov 12. PMID 39531116
- [Derived] Santa Maria DM, Padhye N, Ostrosky-Zeichner L, Grimes CZ, Nyamathi A, Lightfoot M, Quadri Y, Paul ME, Jones JT. COVID-19 Vaccination Uptake, Infection Rates, and Seropositivity Among Youth Experiencing Homelessness in the United States. Nurs Res. 2024 Sep-Oct 01;73(5):373-380. doi: 10.1097/NNR.0000000000000747. Epub 2024 May 10. PMID 38809559

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | NCM4HIV | Usual Care
Started | 318 | 156
Received Intervention | 303 | 147
Completed | 303 | 147
Not Completed | 15 | 9

BASELINE CHARACTERISTICS:
Population: Includes all participants who received intervention.
Groups:
- Total: Total of all reporting groups
Arm/Group | NCM4HIV | Usual Care | Total
Number analyzed (Participants) | 303 | 147 | 450
Age, Continuous [Mean (Standard Deviation); unit: years] | 21 (2.1) | 21.1 (2.1) | 21.1 (2.1)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Female | 138 | 57 | 195
  Male | 149 | 77 | 226
  Transgender Male | 2 | 5 | 7
  Transgender Female | 8 | 3 | 11
  Genderqueer, neither exclusively male nor female | 3 | 2 | 5
  Other | 2 | 2 | 4
  Decline to Answer | 1 | 1 | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 47 | 25 | 72
  Not Hispanic or Latino | 255 | 121 | 376
  Unknown or Not Reported | 1 | 1 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 5 | 0 | 5
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 185 | 94 | 279
  White | 39 | 12 | 51
  More than one race | 37 | 19 | 56
  Unknown or Not Reported | 36 | 22 | 58
Region of Enrollment [Number; unit: participants]
  United States | 303 | 147 | 450

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Use Preventive Prophylaxis (PrEP)
Time Frame: baseline
Measure: Count of Participants; unit: Participants
Arm/Group | NCM4HIV | Usual Care
Number analyzed (Participants) | 303 | 147
Participants | 20 | 18

2. Primary Outcome: Number of Participants Who Use Preventive Prophylaxis (PrEP)
Description: Multiple imputation was used because there were high missing fractions for many variables. This approach assumed that data were missing at random (MAR) and the imputation model used the same multilevel modeling approach that was used for analysis. The models made use of the correlations among repeated measurements for participants to estimate missing values. The descriptive statistics represent averages across 10 imputed data sets.
Time Frame: At completion of the 3-month intervention (Month 3)
Measure: Count of Participants; unit: Participants
Arm/Group | NCM4HIV | Usual Care
Number analyzed (Participants) | 303 | 147
Participants | 55 | 21

3. Primary Outcome: Number of Participants Who Use Preventive Prophylaxis (PrEP)
Description: as for outcome 2
Time Frame: 3 months after intervention (Month 6)
Measure: Count of Participants; unit: Participants
Arm/Group | NCM4HIV | Usual Care
Number analyzed (Participants) | 303 | 147
Participants | 37 | 17

4. Primary Outcome: Number of Participants Who Use Preventive Prophylaxis (PrEP)
Description: as for outcome 2
Time Frame: 6 months after intervention (Month 9)
Measure: Count of Participants; unit: Participants
Arm/Group | NCM4HIV | Usual Care
Number analyzed (Participants) | 303 | 147
Participants | 45 | 17

5. Primary Outcome: Number of Participants Who Use Preventive Prophylaxis (PrEP)
Description: as for outcome 2
Time Frame: 9 months after intervention (Month 12)
Measure: Count of Participants; unit: Participants
Arm/Group | NCM4HIV | Usual Care
Number analyzed (Participants) | 303 | 147
Participants | 42 | 12

6. Primary Outcome: Number of Participants Who Use Non-occupational Post-exposure Prophylaxis (nPEP)
Time Frame: baseline
Measure: Count of Participants; unit: Participants
Arm/Group | NCM4HIV | Usual Care
Number analyzed (Participants) | 303 | 147
Participants | 6 | 14

7. Primary Outcome: Number of Participants Who Use Non-occupational Post-exposure Prophylaxis (nPEP)
Description: as for outcome 2
Time Frame: At completion of the 3-month intervention (Month 3)
Measure: Count of Participants; unit: Participants
Arm/Group | NCM4HIV | Usual Care
Number analyzed (Participants) | 303 | 147
Participants | 7 | 4

8. Primary Outcome: Number of Participants Who Use Non-occupational Post-exposure Prophylaxis (nPEP)
Description: as for outcome 2
Time Frame: 3 months after intervention (Month 6)
Measure: Count of Participants; unit: Participants
Arm/Group | NCM4HIV | Usual Care
Number analyzed (Participants) | 303 | 147
Participants | 6 | 4

9. Primary Outcome: Number of Participants Who Use Non-occupational Post-exposure Prophylaxis (nPEP)
Description: as for outcome 2
Time Frame: 6 months after intervention (Month 9)
Measure: Count of Participants; unit: Participants
Arm/Group | NCM4HIV | Usual Care
Number analyzed (Participants) | 303 | 147
Participants | 10 | 3

10. Primary Outcome: Number of Participants Who Use Non-occupational Post-exposure Prophylaxis (nPEP)
Description: as for outcome 2
Time Frame: 9 months after intervention (Month 12)
Measure: Count of Participants; unit: Participants
Arm/Group | NCM4HIV | Usual Care
Number analyzed (Participants) | 303 | 147
Participants | 6 | 5

11. Primary Outcome: Number of Participants Who Use Condoms at Last Sex as Measured by the Youth Risk Behavior Survey
Description: An item from the Youth Risk Behavior Survey was used to assess this outcome. The items asked if a condom was used at last sex. The number of participants who answered yes is reported.
Time Frame: baseline
Measure: Count of Participants; unit: Participants
Arm/Group | NCM4HIV | Usual Care
Number analyzed (Participants) | 303 | 147
Participants | 86 | 34

12. Primary Outcome: Number of Participants Who Use Condoms at Last Sex as Measured by the Youth Risk Behavior Survey
Description: An item from the Youth Risk Behavior Survey was used to assess this outcome. The items asked if a condom was used at last sex. The number of participants who answered yes is reported.\
  Multiple imputation was used because there were high missing fractions for many variables. This approach assumed that data were missing at random (MAR) and the imputation model used the same multilevel modeling approach that was used for analysis. The models made use of the correlations among repeated measurements for participants to estimate missing values. The descriptive statistics represent averages across 10 imputed data sets.
Time Frame: At completion of the 3-month intervention (Month 3)
Measure: Count of Participants; unit: Participants
Arm/Group | NCM4HIV | Usual Care
Number analyzed (Participants) | 303 | 147
Participants | 81 | 36

13. Primary Outcome: Number of Participants Who Use Condoms at Last Sex as Measured by the Youth Risk Behavior Survey
Description: An item from the Youth Risk Behavior Survey was used to assess this outcome. The items asked if a condom was used at last sex. The number of participants who answered yes is reported.
  Multiple imputation was used because there were high missing fractions for many variables. This approach assumed that data were missing at random (MAR) and the imputation model used the same multilevel modeling approach that was used for analysis. The models made use of the correlations among repeated measurements for participants to estimate missing values. The descriptive statistics represent averages across 10 imputed data sets.
Time Frame: 3 months after intervention (Month 6)
Measure: Count of Participants; unit: Participants
Arm/Group | NCM4HIV | Usual Care
Number analyzed (Participants) | 303 | 147
Participants | 64 | 41

14. Primary Outcome: Number of Participants Who Use Condoms at Last Sex as Measured by the Youth Risk Behavior Survey
Description: as for outcome 13
Time Frame: 6 months after intervention (Month 9)
Measure: Count of Participants; unit: Participants
Arm/Group | NCM4HIV | Usual Care
Number analyzed (Participants) | 303 | 147
Participants | 84 | 23

15. Primary Outcome: Number of Participants Who Use Condoms at Last Sex as Measured by the Youth Risk Behavior Survey
Description: as for outcome 13
Time Frame: 9 months after intervention (Month 12)
Measure: Count of Participants; unit: Participants
Arm/Group | NCM4HIV | Usual Care
Number analyzed (Participants) | 303 | 147
Participants | 74 | 34

16. Primary Outcome: Number of Participants Who Tested Positive for HIV or Sexually Transmitted Infection (STI)
Description: Sexually Transmitted Infection tested includes syphilis, chlamydia and gonorrhea.
Time Frame: Baseline
Measure: Count of Participants; unit: Participants
Arm/Group | NCM4HIV | Usual Care
Number analyzed (Participants) | 303 | 147
Participants | 63 | 24

17. Primary Outcome: Number of Participants Who Tested Positive for HIV or Sexually Transmitted Infection (STI)
Description: Sexually Transmitted Infection tested includes syphilis, chlamydia and gonorrhea.
  Multiple imputation was used because there were high missing fractions for many variables. This approach assumed that data were missing at random (MAR) and the imputation model used the same multilevel modeling approach that was used for analysis. The models made use of the correlations among repeated measurements for participants to estimate missing values. The descriptive statistics represent averages across 10 imputed data sets.
Time Frame: At completion of the 3-month intervention (Month 3)
Measure: Count of Participants; unit: Participants
Arm/Group | NCM4HIV | Usual Care
Number analyzed (Participants) | 303 | 147
Participants | 43 | 19

18. Primary Outcome: Number of Participants Who Tested Positive for HIV or Sexually Transmitted Infection (STI)
Description: as for outcome 17
Time Frame: 3 months after intervention (Month 6)
Measure: Count of Participants; unit: Participants
Arm/Group | NCM4HIV | Usual Care
Number analyzed (Participants) | 303 | 147
Participants | 32 | 13

19. Primary Outcome: Number of Participants Who Tested Positive for HIV or Sexually Transmitted Infection (STI)
Description: as for outcome 17
Time Frame: 6 months after intervention (Month 9)
Measure: Count of Participants; unit: Participants
Arm/Group | NCM4HIV | Usual Care
Number analyzed (Participants) | 303 | 147
Participants | 44 | 24

20. Primary Outcome: Number of Participants Who Tested Positive for HIV or Sexually Transmitted Infection (STI)
Description: as for outcome 17
Time Frame: 9 months after intervention (Month 12)
Measure: Count of Participants; unit: Participants
Arm/Group | NCM4HIV | Usual Care
Number analyzed (Participants) | 303 | 147
Participants | 38 | 18

21. Secondary Outcome: Mental Health as Measured by the Brief Symptom Index-18
Description: The Brief Symptom Inventory 18 (BSI-18) consists of 18 items on a 5-point (0-4) Likert scale and is designed to assess current psychological distress (over the past 7 days). Total score ranges from 0 to 72, with higher scores indicating greater distress.
Time Frame: baseline
Population: Data were not collected for this outcome measure because the Brief Symptom Index-18 survey was not administered to participants. Instead, the Patient Health Questionnaire (PHQ-9) was used to assess mental health. As a result, no participants received the Brief Symptom Index-18 survey, and no data were collected for this outcome measure. Therefore, zero participants were analyzed for this outcome. Data from the PHQ-9 are reported under a different outcome measure.
Arm/Group | NCM4HIV | Usual Care
Number analyzed (Participants) | 0 | 0

22. Secondary Outcome: Mental Health as Measured by the Brief Symptom Index-18
Description: The BSI-18 consists of 18 items on a 5-point (0-4) Likert scale and is designed to assess current psychological distress (over the past 7 days). Total score ranges from 0 to 72, with higher scores indicating greater distress.
Time Frame: At completion of the 3-month intervention (Month 3)
Population: as for outcome 21
Arm/Group | NCM4HIV | Usual Care
Number analyzed (Participants) | 0 | 0

23. Secondary Outcome: Mental Health as Measured by the Brief Symptom Index-18
Description: as for outcome 22
Time Frame: 3 months after intervention (Month 6)
Population: as for outcome 21
Arm/Group | NCM4HIV | Usual Care
Number analyzed (Participants) | 0 | 0

24. Secondary Outcome: Mental Health as Measured by the Brief Symptom Index-18
Description: as for outcome 22
Time Frame: 6 months after intervention (Month 9)
Population: as for outcome 21
Arm/Group | NCM4HIV | Usual Care
Number analyzed (Participants) | 0 | 0

25. Secondary Outcome: Mental Health as Measured by the Brief Symptom Index-18
Description: as for outcome 22
Time Frame: 9 months after intervention (Month 12)
Population: as for outcome 21
Arm/Group | NCM4HIV | Usual Care
Number analyzed (Participants) | 0 | 0

26. Secondary Outcome: Housing Status
Description: Participants will be asked if they live in a shelter, apartment/house, with someone, outside, or in a car, etc.
Time Frame: baseline
Measure: Count of Participants; unit: Participants
Arm/Group | NCM4HIV | Usual Care
Number analyzed (Participants) | 303 | 147
Participants
  My own place | 13 | 7
  Family/Foster Family home | 16 | 2
  Friend's home | 41 | 14
  Home of boyfriend/girlfriend/sexual partner | 4 | 1
  Shelter | 181 | 95
  Hotel or motel | 2 | 3
  Transitional living program | 10 | 5
  street, park, or outside | 17 | 10
  abandoned building or squat | 9 | 4
  car, bus, light rail, or metro | 2 | 1
  Other | 7 | 5
  Unknown/Not Reported | 1 | 0

27. Secondary Outcome: Housing Status
Description: Participants will be asked if they live in a shelter, apartment/house, with someone, outside, or in a car, etc.
Time Frame: At completion of the 3-month intervention (Month 3)
Population: Data were not collected for 82 participants in the NCM4HIV arm and 39 participants in the Usual Care arm due to loss to follow-up
Measure: Count of Participants; unit: Participants
Arm/Group | NCM4HIV | Usual Care
Number analyzed (Participants) | 221 | 108
Participants
  My own place | 33 | 16
  Family/Foster Family Home | 25 | 8
  Friend's Home | 24 | 14
  Home of boyfriend/girlfriend/sexual partner | 5 | 6
  Shelter | 103 | 46
  Hotel or Motel | 8 | 5
  Transitional living program | 9 | 5
  Street, park or outside | 8 | 4
  Abandoned building or squat | 3 | 0
  car, bus, light rail, or metro | 1 | 1
  Other | 2 | 3

28. Secondary Outcome: Housing Status
Description: Participants will be asked if they live in a shelter, apartment/house, with someone, outside, or in a car, etc.
Time Frame: 3 months after intervention (Month 6)
Population: Data were not collected for 117 participants in the NCM4HIV arm and 62 participants in the Usual Care arm due to loss to follow-up
Measure: Count of Participants; unit: Participants
Arm/Group | NCM4HIV | Usual Care
Number analyzed (Participants) | 186 | 85
Participants
  My own place | 49 | 15
  Family/Foster Family home | 21 | 12
  Friend's home | 21 | 14
  Home of boyfriend/girlfriend/sexual partner | 8 | 6
  Shelter | 60 | 17
  Hotel or motel | 8 | 4
  Transitional living program | 3 | 4
  street, park, or outside | 6 | 6
  abandoned building or squat | 3 | 0
  car, bus, light rail, or metro | 0 | 3
  Other | 7 | 4

29. Secondary Outcome: Housing Status
Description: Participants will be asked if they live in a shelter, apartment/house, with someone, outside, or in a car, etc.
Time Frame: 6 months after intervention (Month 9)
Population: Data were not collected for 129 participants in the NCM4HIV arm and 71 participants in the Usual Care arm due to loss to follow-up
Measure: Count of Participants; unit: Participants
Arm/Group | NCM4HIV | Usual Care
Number analyzed (Participants) | 174 | 76
Participants
  My own place | 64 | 18
  Family/Foster Family home | 17 | 13
  Friend's home | 23 | 8
  Home of boyfriend/girlfriend/sexual partner | 8 | 3
  Shelter | 33 | 19
  Hotel or motel | 10 | 5
  Transitional living program | 3 | 2
  street, park, or outside | 5 | 5
  abandoned building or squat | 3 | 1
  car, bus, light rail, or metro | 2 | 0
  Other | 6 | 2

30. Secondary Outcome: Housing Status
Description: Participants will be asked if they live in a shelter, apartment/house, with someone, outside, or in a car, etc.
Time Frame: 9 months after intervention (Month 12)
Population: Data were not collected for 119 participants in the NCM4HIV arm and 65 participants in the Usual Care arm due to loss to follow-up
Measure: Count of Participants; unit: Participants
Arm/Group | NCM4HIV | Usual Care
Number analyzed (Participants) | 184 | 82
Participants
  My own place | 69 | 23
  Family/Foster Family home | 27 | 14
  Friend's home | 19 | 13
  Home of boyfriend/girlfriend/sexual partner | 12 | 2
  Shelter | 21 | 12
  Hotel or motel | 7 | 2
  Transitional living program | 5 | 1
  street, park, or outside | 9 | 7
  abandoned building or squat | 2 | 1
  car, bus, light rail, or metro | 5 | 2
  Other | 8 | 5

31. Secondary Outcome: Number of Participants With Substance Use as Measured by Item 11 in the Texas Christian University (TCU) Drug Screen II
Description: An item from the Texas Christian University (TCU) drug screen II was used to assess this outcome. The item listed various drug substances and asked whether any of those listed had been used in the past 30 days. The number of participants who answered yes is reported.
  Multiple imputation was used because there were high missing fractions for many variables. This approach assumed that data were missing at random (MAR) and the imputation model used the same multilevel modeling approach that was used for analysis. The models made use of the correlations among repeated measurements for participants to estimate missing values. The descriptive statistics represent averages across 10 imputed data sets.
Time Frame: At completion of the 3-month intervention (Month 3), 3 months after intervention (Month 6), 6 months after intervention (Month 9), 9 months after intervention (Month 12)
Measure: Count of Participants; unit: Participants
Arm/Group | NCM4HIV | Usual Care
Number analyzed (Participants) | 303 | 147
Participants
  At completion of the 3-month intervention (Month 3) | 162 | 70
  3 months after intervention (Month 6) | 140 | 79
  6 months after intervention (Month 9) | 138 | 74
  9 months after intervention (Month 12) | 146 | 60

32. Secondary Outcome: Mental Health as Measured by the Patient Health Questionnaire (PHQ-9)
Description: The Patient Health Questionnaire (PHQ-9) total score ranges from 0 to 27, with higher scores indicating more severe depression
Time Frame: baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | NCM4HIV | Usual Care
Number analyzed (Participants) | 303 | 147
score on a scale | 8.8 (6.99) | 8.5 (7.25)

33. Secondary Outcome: Mental Health as Measured by the Patient Health Questionnaire (PHQ-9)
Description: The Patient Health Questionnaire (PHQ-9) total score ranges from 0 to 27, with higher scores indicating more severe depression.
  Multiple imputation was used because there were high missing fractions for many variables. This approach assumed that data were missing at random (MAR) and the imputation model used the same multilevel modeling approach that was used for analysis. The models made use of the correlations among repeated measurements for participants to estimate missing values. The descriptive statistics represent averages across 10 imputed data sets.
Time Frame: At completion of the 3-month intervention (Month 3)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | NCM4HIV | Usual Care
Number analyzed (Participants) | 303 | 147
score on a scale | 7.7 (6.81) | 8.9 (7.92)

34. Secondary Outcome: Mental Health as Measured by the Patient Health Questionnaire (PHQ-9)
Description: as for outcome 33
Time Frame: 3 months after intervention (Month 6)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | NCM4HIV | Usual Care
Number analyzed (Participants) | 303 | 147
score on a scale | 6.9 (6.82) | 8.1 (7.52)

35. Secondary Outcome: Mental Health as Measured by the Patient Health Questionnaire (PHQ-9)
Description: as for outcome 33
Time Frame: 6 months after intervention (Month 9)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | NCM4HIV | Usual Care
Number analyzed (Participants) | 303 | 147
score on a scale | 7.3 (7.09) | 8 (7.21)

36. Secondary Outcome: Mental Health as Measured by the Patient Health Questionnaire (PHQ-9)
Description: as for outcome 33
Time Frame: 9 months after intervention (Month 12)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | NCM4HIV | Usual Care
Number analyzed (Participants) | 303 | 147
score on a scale | 7.7 (7.09) | 6.6 (6.73)

37. Secondary Outcome: Number of Participants With Substance Use as Measured by Item 11 in the Texas Christian University (TCU) Drug Screen II
Description: An item from the Texas Christian University (TCU) drug screen II was used to assess this outcome. The item listed various drug substances and asked whether any of those listed had been used in the past 30 days. The number of participants who answered yes is reported.
Time Frame: baseline
Measure: Count of Participants; unit: Participants
Arm/Group | NCM4HIV | Usual Care
Number analyzed (Participants) | 303 | 147
Participants | 170 | 79

ADVERSE EVENTS:
Time Frame: up to 1 year
Arm/Group | NCM4HIV | Usual Care
All-Cause Mortality (participants affected / at risk) | 1/318 | 2/156
Serious Adverse Events (participants affected / at risk) | 5/318 | 1/156
Other Adverse Events (participants affected / at risk) | 0/318 | 0/156
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | NCM4HIV (N=318) | Usual Care (N=156)
Suicidal ideation (Psychiatric disorders) | 1 (2) | 1 (1)
Hospitalization (General disorders) | 1 (1) | 0 (0)
Hospitalization (Psychiatric disorders) | 2 (2) | 0 (0)
Reported child abuse (General disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-03-09): https://cdn.clinicaltrials.gov/large-docs/18/NCT03910218/Prot_SAP_000.pdf
  • Informed Consent Form (2021-03-09): https://cdn.clinicaltrials.gov/large-docs/18/NCT03910218/ICF_001.pdf